CLINICAL TRIAL: NCT00528008
Title: Povidone-iodine vs. Chlorhexidine Gluconate - A Comparison of Surgical Preparations and Wound Infection Rates for Elective Cesarean Sections
Brief Title: A Comparison of Surgical Preparations and Wound Infection Rates for Elective Cesarean Sections
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study was stopped following interim analysis.
Sponsor: Memorial University of Newfoundland (Other)
Collaborators: Eastern Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HIC07.33
Record Dates: First submitted 2007-09-10; First posted 2007-09-11 (Estimated); Last update posted 2012-11-09 (Estimated); Status verified 2012-11

CONDITIONS: Wound Infection
Keywords: infection; sepsis; povidone-iodine; chlorhexidine gluconate; fever; erythema; leukocytosis; drainage; vaginal discharge; elective cesarean section
MeSH Terms: conditions — Wound Infection; Infections; Sepsis; Fever; Erythema; Leukocytosis; Vaginal Discharge | interventions — Povidone-Iodine; Povidone; chlorhexidine gluconate; Chlorhexidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): povidone-iodine
  Interventions: Other: povidone-iodine solution
- B (Active Comparator): chlorhexidine gluconate
  Interventions: Other: chlorhexidine gluconate

INTERVENTIONS:
Other: povidone-iodine solution — Abdominal surgical field cleaned with 5% povidone-iodine detergent scrub, detergent cleaned from surgical area with sterile water, and then painted with 1% povidone-iodine solution.
  Other Names: Betadine, Povidone, Minidyne
  Arms: A
Other: chlorhexidine gluconate — Abdominal surgical field painted once using 2% chlorhexidine in 70% alcohol.
  Other Names: Dexidine, Avagard, Bactoshield
  Arms: B

SUMMARY:
The purpose of this study is to find out if chlorhexidine gluconate solution is better at reducing the rate of wound infection after cesarean section compared to povidone-iodine.

DETAILED DESCRIPTION:
Wound infection is a universal potential morbidity to any type of surgery. Over the years many studies have been completed to evaluate ways to decrease this morbidity. Recent literature has looked at different types of surgical solutions used in pre-operative cleansing. Chlorhexidine and povidone-iodine are two standard surgical prep solutions used on a global scale. The most recent literature has shown that chlorhexidine has a decreased wound infection rate for longer surgeries. Cesarean section, as a surgical time, varies from 20 - 60 minutes. There has been no known literature regarding wound infection rates using these two solutions in elective cesarean sections. This trial will review the rates of wound infection using chlorhexidine and povidone-iodine during elective cesarean section and determine if there is any statistically significant difference between the two solutions. The results could potentially decrease wound infection rates, decrease morbidity, decrease hospital length of stay, and help to guide further surgical management.

ELIGIBILITY:
Inclusion Criteria:

* Age >19 years
* Gestational age > 37 weeks
* Booked elective cesarean section

Exclusion Criteria:

* Gestational age < 37 weeks
* Premature rupture of membranes
* Onset of labor prior to procedure
* Evidence of maternal sepsis; maternal fever > 38.5C
* LSCS for emergency issues: non-reassuring fetal status, placental abruption, failed induction

Min Age: 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 268 (Actual)
Dates: Start 2007-12; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
to determine the rate of wound infection using two standard wound preparations: povidone-iodine and chlorhexidine gluconate | within 6 weeks following surgery

SECONDARY OUTCOMES:
readmission to hospital | within 6 weeks following surgery
extended length of admission | within 6 weeks following surgery
need for intravenous antibiotics | within 6 weeks following surgery
need for repeat procedure such as drainage | within 6 weeks following surgery
increased outpatient surveillance | within 6 weeks following surgery

CONTACTS AND LOCATIONS:
Overall Officials: Paula Mallaley, MD, Principal Investigator — Resident, Obstetrics and Gynecology, Memorial University of Newfoundland
Locations (1):
- Women' s Health Centre, Eastern Health, St. John's, Newfoundland and Labrador, Canada